CLINICAL TRIAL: NCT00734526
Title: A Phase I Study of Sorafenib With Radiation and Temozolomide in Newly Diagnosed Glioblastoma or Gliosarcoma
Brief Title: Phase I Portion of Phase I/II Sorafenib With Radiation and Temozolomide in Newly Diagnosed Glioblastoma or Gliosarcoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0059; NCI-2012-01617 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Glioblastoma; Gliosarcoma
Keywords: Glioblastoma; Gliosarcoma; Brain Cancer; Sorafenib; Temozolomide; Radiation; Radiotherapy; XRT
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — Temozolomide; Radiation; Radiotherapy; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dose Level 1 (Experimental): Temozolomide + Radiation, Followed by Higher Dose Temozolomide in a Shorter Cycle
  Temozolomide 75mg/m^2 daily during radiation therapy, and 150mg/m^2 in the first cycle of adjuvant therapy. Dose Level 1 will receive sorafenib in the adjuvant phase (following radiation therapy) at the dose of 400mg BID in combination with standard dose temozolomide 150-200 mg/m^2 two days out of 28 day cycle. Radiotherapy 2.0 Grey (Gy)/day given daily 5 days per week for total of 60.0 Gy over 6 weeks.
  Interventions: Drug: Temozolomide; Radiation: Radiation; Drug: Sorafenib
- 2 (Experimental): Temozolomide + Lower Dose Sorafenib + Radiation, Followed by Higher Dose Temozolomide in a Shorter Cycle + Higher Dose Sorafenib
  Interventions: Drug: Temozolomide; Radiation: Radiation; Drug: Sorafenib
- 3 (Experimental): Temozolomide + Lower Dose Sorafenib + Radiation, Followed by Lower Dose Temozolomide in a Longer Cycle + Lower Dose Sorafenib
  Interventions: Drug: Temozolomide; Radiation: Radiation; Drug: Sorafenib
- 4 (Experimental): Temozolomide + Higher Dose Sorafenib + Radiation, Followed by Lower Dose Temozolomide in a Longer Cycle + Higher Dose Sorafenib
  Interventions: Drug: Temozolomide; Radiation: Radiation; Drug: Sorafenib

INTERVENTIONS:
Drug: Temozolomide — Groups 1 & 2: 75 mg/m^2 Once Daily by Mouth During Radiation; 4 Weeks after Completion of Radiation, 150-200 mg/m^2 Once Daily by Mouth Days 1-5 of 1st 28-Day Cycle, then 75 mg/m^2 Once Daily by Mouth Days 1-5 for Subsequent 28-Day Cycles.
  Groups 3 & 4: 75 mg/m^2 Once Daily by Mouth During Radiation; 4 Weeks after Completion of Radiation, 75-100 mg/m^2 Once Daily by Mouth Days 1-21 every 28-Day Cycle.
Radiation: Radiation — Total of 60 Gy delivered over 30 Days (approximately 6 weeks).
  Other Names: Radiotherapy; XRT
Drug: Sorafenib — Group 1: 4 Weeks after Completion of Radiation, 400 mg Twice Daily by Mouth.
  Group 2: 200 mg Twice Daily by Mouth during Radiation; 4 Weeks after Completion of Radiation, 400 mg Twice Daily by Mouth.
  Group 3: 200 mg Twice Daily by Mouth during Radiation; 4 Weeks after Completion of Radiation, 200 mg Twice Daily by Mouth.
  Group 4: 400 mg Twice Daily by Mouth during Radiation; 4 Weeks after Completion of Radiation, 400 mg Twice Daily by Mouth.
  Other Names: BAY43-9006

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of sorafenib that can be given in combination with temozolomide. The safety of this combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Sorafenib is designed to stop the cell growth and to block the formation of new blood vessels (the tubes that carry blood around the body), which are involved in the growth and development of tumors.

Temozolomide is designed to kill cancer cells by damaging DNA (the genetic material of cells). The damaged DNA may cause tumor cell death.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to 1 of 4 groups based on when you joined this study. You will remain in the same group for the entire study. In this study, the dose of the study drugs is different from group to group, and the doses are also different during and after radiation. During radiation, the study drugs and doses are as follows:

* If you are in Group 1, you will take temozolomide.
* If you are in Groups 2 or 3, you will take temozolomide and the lower dose of sorafenib.
* If you are in Group 4, you will take temozolomide and the higher dose of sorafenib.
* During radiation, all the groups will take the same dose of temozolomide.

After Radiation:

* If you are in Groups 1 or 2, you will take the higher dose of temozolomide on a shorter cycle and the higher dose of sorafenib.
* If you are in Group 3, you will take the lower dose of temozolomide on a longer cycle and the lower dose of sorafenib.
* If you are in Group 4, you will take the lower dose of temozolomide on a longer cycle and the higher dose of sorafenib.

The amount of study drugs you receive may change if you experience side effects. If at any time you experience any intolerable side effects, tell the study doctor right away.

Study Drug Administration:

During Radiation:

As a part of standard of care, you will receive radiation therapy Monday-Friday for a total of 30 radiation treatments (about 6 weeks).

Every day while you are receiving radiation, you will take the temozolomide by mouth once a day (up to a maximum of 7 weeks). On Monday-Friday, you will take temozolomide 1 hour before radiation therapy. On Saturday and Sunday, you will take temozolomide in the morning.

You should swallow temozolomide whole, one right after the other, without chewing them. If you vomit while taking temozolomide, you cannot take more capsules before the next scheduled dose. They should be taken on an empty stomach (at least 1 hour before and 2 hours after eating) with 1 cup (about 8 oz.) of water.

Every day while you are receiving radiation, you will take sorafenib by mouth 2 times a day (in the morning and evening) (up to a maximum of 7 weeks). You should take sorafenib without food (1 hour before or 2 hours after eating), with at least 1 cup (8 oz.) of water. If you are in Group 1, you will not take sorafenib.

After Radiation:

You will not take the study drug(s) for about 4 weeks after the radiation therapy ends.

After 4 weeks:

* If you are in Group 1 or 2, on Days 1-5 of every 28-day study cycle, you will take temozolomide by mouth once a day.
* If you are in Group 3 or 4, on Days 1-21 of every cycle, you will take temozolomide by mouth once a day.

Every day of each cycle, all groups will take sorafenib by mouth 2 times (in the morning and evening).

Study Visits:

During Radiation:

Once a week while you are receiving radiation therapy, you will be asked about any drugs you may be taking and if you have experienced any side effects. Your blood pressure will be measured. Blood (about 3-4 teaspoons) will be drawn for routine tests.

After Radiation:

About 3-4 weeks after the end of radiation therapy, you will have a MRI scan to check the status of the disease.

On Day 1 of every cycle, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs.
* You will have a neurological exam.
* You will have a performance status evaluation.
* You will be asked about any drugs you may be taking and if you have experienced any side effects.
* Blood (about 3-4 teaspoons) will be drawn for routine tests.

On Days 7, 14, and 21 of Cycle 1 and on Days 7 and 14 (or 21) of Cycles 2 and beyond, blood (about 3-4 teaspoons) will be drawn for routine tests.

On Day 1 of every other cycle (Cycles 3, 5, 7, and so on), you will have a MRI scan to check the status of the disease.

Every week of Cycle 1, your blood pressure will be measured.

Length of Study:

You will be on study for about 15 months total. You will be taken off study early if the disease gets worse or you experience intolerable side effects.

End-of-Study Visit:

After you go off study, you will have an end-of-study visit. At this visit, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your weight and vital signs.
* You will be have a performance status evaluation.
* You will be asked about any drugs you may be taking and if you have experienced any side effects.
* You will have a neurological exam.
* You will have a MRI scan to check the status of the disease.
* Blood (about 3 teaspoons) will be drawn for routine tests.

This is an investigational study. Temozolomide is FDA approved and commercially available for the treatment of brain tumors. Sorafenib is FDA approved and commercially available for the treatment of kidney cancer, but it is experimental for use in brain tumors. In addition, the combination of temozolomide and Sorafenib is experimental for use in brain tumors. At this time, the combination is only being used in research.

Up to 51 participants will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically proven diagnosis of glioblastoma. Since gliosarcoma is a variant of glioblastoma, gliosarcoma is also an eligible diagnosis.
2. Patients must have at least 1 block of tumor tissue available for submission to the central pathologist for analysis of gene expression status by QRT-PCR; there must be at least 1 cm^2 of tumor from the block when cut on a slide: fresh frozen tumor tissue acquisition is also encouraged, but not required. Unstained slide submission without a block submission is not acceptable for study entry.
3. Diagnosis must be established by open biopsy or tumor resection. Patients who have only had a stereotactic biopsy are not eligible..
4. The tumor must have a supratentorial component.
5. Patients must have recovered from the effects of surgery, postoperative infection, and other complications before study registration.
6. All patients must sign an informed consent indicating that they are aware of the investigational nature of this study.
7. A diagnostic contrast-enhanced MRI or CT scan (if MRI is contraindicated) of the brain must be performed postoperatively in the period between surgery and initiation of radiation therapy.
8. Therapy must begin </=5 weeks after the most recent brain tumor surgery.
9. History/physical examination within 14 days prior to study registration.
10. Neurologic examination within 14 days prior to study registration.
11. Documentation of steroid doses within 14 days prior to study registration and stable or decreasing steroid dose within 5 days prior to registration.
12. Karnofsky performance status of >/= 60.
13. Age >/= 18 years.
14. Patients with well-controlled hypertension are eligible (systolic blood pressure of </= 140 mgHg or diastolic pressure </= 90 mgHg).
15. Complete blood count (CBC)/differential obtained within 14 days prior to study registration, with adequate bone marrow function as defined below: Absolute neutrophil count (ANC) >/= 1500 cells/mm^3; Platelets >/= 100,000 cells/mm^3;Hemoglobin >/= 10 g/dl.
16. Adequate renal function, as defined below: Serum creatinine </= 1.7 mg/dl within 14 days prior to study registration
17. Adequate hepatic function, as defined below: Bilirubin </= 2.0 mg/dl within 14 days prior to study registration; ALT </= 2 x upper limit of normal range (ULN) within 14 days prior to study registration; AST </= 2 x ULN range within 14 days prior to study registration
18. Fasting cholesterol < 300 mg/dL (9.0 mmol/L) and fasting triglycerides < 2.5 times ULN
19. International normalized ratio (INR) < 1.5 or a PT/PTT within normal limits for patients not on anti-coagulation treatment
20. Patients receiving anti-coagulation treatment with an agent such as warfarin or low molecular weight heparin may be allowed to participate with the following criteria: For patients on prophylactic anticoagulation therapy (low-dose warfarin): INR level < 1.5; Patients on prophylactic dose or full dose low molecular weight heparins are eligible provided that the patient has no active bleeding or pathological condition that carries a high risk of bleeding;
21. (20. continued) Patients on full-dose anticoagulants (e.g., warfarin) are eligible provided that both of the following criteria are met: (a) Patient has an in-range INR (usually between 2-3) on a stable dose or oral anticoagulant or on a stable dose of low molecular weight heparin. (b) Patient has no active bleeding or pathological condition that carries a high risk of bleeding.
22. If the patient's mental status precludes his/her giving informed consent, written informed consent may be given by the responsible family member.
23. For females of child-bearing potential, negative serum pregnancy test within 72 hours prior to starting temozolomide
24. Women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation. Men should use adequate birth control for at least six months after the last administration of sorafenib or temozolomide.

Exclusion Criteria:

1. Prior invasive malignancy (except for non-melanomatous skin cancer) unless disease free for >/= 3 years.
2. Recurrent or multifocal malignant gliomas
3. Metastases detected below the tentorium or beyond the cranial vault.
4. Prior chemotherapy or radiosensitizers for cancers of the head and neck region; note that prior chemotherapy for a different cancer is allowable.
5. Prior use of Gliadel wafers or any other intratumoral or intracavitary treatment are not permitted.
6. Prior radiotherapy to the head or neck (except for T1 glottic cancer), resulting in overlap of radiation fields.
7. Severe, active co-morbidity, defined as follows: Cardiac disease - Congestive heart failure > class II New York Heart Association (NYHA). Patients must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months; Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy; Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration; Chronic Hepatitis B or C infection;
8. (7. continued) Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration; Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects;
9. (7. continued) Known history or symptoms and laboratory results consistent with Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition (note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive); Major medical illnesses or psychiatric impairments that in the investigator's opinion will prevent administration or completion of protocol therapy;
10. (7. continued) Active connective tissue disorders, such as lupus or scleroderma, that in the opinion of the treating physician may put the patient at high risk for radiation toxicity; Arterial thrombotic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months; Pulmonary hemorrhage/bleeding event > Common Toxicity Criteria for Adverse Effects (CTCAE) Grade 2 within 4 weeks of first dose of study drug;
11. (7. continued) Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug; Serious non-healing wound, ulcer, or bone fracture; Evidence or history of bleeding diathesis or coagulopathy
12. Uncontrolled hypertension defined as systolic blood pressure > 140 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.
13. Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study drug.
14. Use of St. John's Wort or rifampin (rifampicin).
15. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.
16. No tissue provided for histopathologic review and QRT-PCR analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-12-18 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Phase I: Sorafenib Maximum Tolerated Dose (MTD) | 4 Week Cycles
  MTD of sorafenib given during (concurrently with) external beam radiation therapy and daily temozolomide (75mg/m^2), and with standard dose temozolomide (150-200mg/m^2 5 days out of 28) after radiation therapy (adjuvant) in patients with newly diagnosed glioblastoma or gliosarcoma
  MTD is defined as the dose level below which there were 2 or more participants out of 6 with Dose-limiting toxicities (DLTs). by the conclusion of the first cycle of post-radiation therapy (14 weeks),
Second MTD | 4 weeks
  maximum tolerated dose (MTD) of sorafenib given during (concurrently with) external beam radiation therapy and daily temozolomide (75mg/m2), and with dose dense temozolomide (100mg/m2 21 days out of 28) after radiation therapy (adjuvant) in patients with newly diagnosed glioblastoma or gliosarcoma

SECONDARY OUTCOMES:
Phase II: Time to Progression | 15 Months or till progressive disease, severe toxicity or death.

CONTACTS AND LOCATIONS:
Overall Officials: Vinay K. Puduvalli, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org